CLINICAL TRIAL: NCT05106673
Title: Clinical Implementation and Evaluation of Three Implementation Interventions for a Family-oriented Care for Children of Mentally Ill Parents (Ci-CHIMPS)
Brief Title: Clinical Implementation and Evaluation for the Family-oriented Care CHIMPS-NET
Acronym: Ci-Chimps
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: Evangelisches Klinikum Bethel (Unknown); Charite University, Berlin, Germany (Other); Universitätsklinikum Leipzig (Other); University Hospital, Saarland (Other); Immanuel Klinik Rüdersdorf (Unknown); LWL Klinik Gütersloh (Unknown); University Hospital, Aachen (Other); University of Ulm (Other); Universitätsklinikum Köln (Other); University Hospital Freiburg (Other); University Hospital Augsburg (Other); University Medical Center Rostock (Other); University Hospital Tuebingen (Other); Helios Kliniken Schwerin (Other); University of Magdeburg (Other); Universitätsklinikum Koblenz - Landau (Unknown); HELIOS Hospital, Erfurt, Germany (Other); Goethe University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Ci-Chimps
Record Dates: First submitted 2021-10-24; First posted 2021-11-04 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: Mental Health Issue
Keywords: Children of mentally ill parents; implementation research; family implementation interventions; Randomized controlled trial
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: The study will include two groups: one intervention group (IG) and one control group (TAU). The intervention group includes three different interventions.
Masking Description: There is no masking.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- clinical centers that receive implementation support (Experimental): These clinical centers receive support during the implementation of the CHIMPS-intervention. There are three different implementation interventions.
  Interventions: Behavioral: Optimal pathways to care; Behavioral: Education and training program for the professionals; Behavioral: Systematic screening
- No Intervention: Treatment as usual (Experimental): These clinical centers will be the control group and will not get a specific implementation support during the implementation of CHIMPS.
  Interventions: Other: TAU

INTERVENTIONS:
Behavioral: Optimal pathways to care — The first implementation measure focuses on optimal ways of caring for mentally ill patients who are also parents with children living in the household. The main goals of this intervention are the specific information of the referring physician, the indicated referral of mentally ill parents and the consideration of underage children living in the household in the inpatient referral. The two main components are the evaluation of the attitudes of the medical and psychotherapeutic referrers towards the target group and the intervention as well as the development and implementation of an optimal care pathway. The optimization of the allocation is organized by Silke Pawils (University Medical Center Hamburg-Eppendorf).
  Arms: clinical centers that receive implementation support
Behavioral: Education and training program for the professionals — The second implementation intervention concerns the improvement of the professionals' attitudes, knowledge and skills. The two main components here being the assessment of the current state in all institutions within the clinical centers and the development and implementation of an education and training program. The employees of the randomized clinical centers in the intervention group will get a three-hour training. This intervention is organized by Svenja Taubner (University Hospital Heidelberg, Germany).
  Arms: clinical centers that receive implementation support
Behavioral: Systematic screening — The third implementation intervention includes a systematic screening process to improve detection of mentally ill parents with affected children. Employees of the clinical centers fill out two short questionnaires with the parents. This intervention project is organized by Sibylle M. Winter (Charité, Berlin, Germany).
  Arms: clinical centers that receive implementation support
Other: TAU — No Intervention: Treatment as usual These clinical centers will be the control group and will not get a specific implementation support during the implementation of CHIMPS.
  Arms: No Intervention: Treatment as usual

SUMMARY:
Despite the knowledge, that children of mentally ill parents are an important target group to be addressed by preventive and therapeutical interventions, there is often a lack of structured implementation of family-oriented interventions in clinical practice in Germany. Using a randomized controlled multicenter trial design with a large and wide-ranging sample (clinics for adult psychiatry and clinics for child and adolescent psychiatry, university clinics and clinics at the real health care) will examine changes in family-oriented practice and aspects of implementation to get a robust understanding of implementing family-oriented interventions in German clinical practice.

DETAILED DESCRIPTION:
A two-group randomized controlled multicenter trial will examine changes in family-oriented practice and aspects of implementation at baseline as well as at 12- and 24-months follow-up. The CHIMPS-Network consists of twenty clinical centers. The centers in the intervention group receive the support of all of the three implementation interventions: 1) Optimal pathways to care 2) Education and a training program for professionals and 3) Systematic screening for children. The centers in the control group do not get this specific implementation support.

The implementation of all the CHIMPS interventions refers to and builds on a theoretical model developed by researchers from Australia and Norway, adapted to the German care system setting including adult psychiatry and child and adolescent psychiatry.

In ci-CHIMPS we aim to determine if three implementation interventions are helpful in improving the clinical implementation of the CHIMPS-NET interventions. Additionally, we want to identify factors hindering or promoting implementation processes. In order to monitor the impact of the three implementation interventions we will use the translated version of the "Family Focused Mental Health Practice Questionnaire (FFMHPQ)" (Laser et al., 2019, in prep.) and the translated version of the "Implementation Components Questionnaire (ICQ)" (Laser, Skogøy, Maybery & Wiegand-Grefe, 2019. in prep). The introduction of these questionnaires in Germany has not yet been reported.

ELIGIBILITY:
Inclusion Criteria:

* Every employee, which is involved in the treatment of the patients (Medicine, Psychology, Nurses) of every clinical center that is part of the CHIMPS-NET project will be invited to participate in this study ci-CHIMPS.

Exclusion Criteria:

* There are no explicit criteria for exclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 798 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Family Focused Mental Health Practice Questionnaire (FFMHPQ) | Change from baseline of the study at 12- and 24-months follow-up
  Measures numerous aspects relevant for family-oriented practice from the employee's point of view with the translated version of the 'Family Focused Mental Health Practice Questionnaire (FFMHPQ)'. (Laser C, Reupert A, Wiegand-Grefe S, Maybery D. Fragebogen zur familienorientierten Arbeit im psychosozialen Gesundheitswesen - deutsche Übersetzung des "Family Focused Mental Health Practice" von Maybery, Goodyear & Reupert. 2019. (in prep.)
Implementation Components Questionnaire (ICQ-35) | Change from baseline of the study at 12- and 24-months follow-up
  Measures from the employee's point of view their perceived level of integration of the intervention within their clinical center. It determines special components of implementation with the translated version of the 'Implementation Components Questionnaire (ICQ-35)'. (Laser, Skogøy, Maybery & Wiegand-Grefe. Implementierungs-Komponenten-Fragebogen.2019. (in prep.)
Implementation Satisfaction Scale (ISS) | Change from baseline of the study at 12- and 24-months follow-up
  Measures from the employee's point of view how satisfied they are with the implementation process in their clinical centre. (Laser, Skogøy, Maybery & Wiegand-Grefe. Implementierungs-Komponenten-Fragebogen.2019. (in prep.)

SECONDARY OUTCOMES:
Sociodemografic information | At baseline of the study
  Sociodemografic information of the employees, assessed from the perspective of the employees

CONTACTS AND LOCATIONS:
Overall Officials: Silke Wiegand-Grefe, Prof. Dr., Study Director — Universitätsklinikum Hamburg-Eppendorf
Locations (1):
- Universitätsklinikum Hamburg Eppendorf, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known if there will be a plan to make IPD available.

REFERENCES:
- [Derived] Laser C, Pawils S, Daubmann A, Zapf A, Wiegand-Grefe S. Different perspectives in psychiatry: how family-oriented are professionals in Germany? BMC Psychiatry. 2024 Feb 20;24(1):142. doi: 10.1186/s12888-024-05562-0. PMID 38378503